CLINICAL TRIAL: NCT07232940
Title: Comparison of the Effects of Ultrasound-Guided Erector Spinae Plane Block and Serratus Posterior Superior Intercostal Plane Block on Postoperative Analgesia Management in Patients Undergoing Video-Assisted Thoracoscopic Surgery
Brief Title: ESP vs SPSIP Block in VATS Analgesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Collaborators: Emre ULUSOY (Unknown)
Responsible Party: Principal Investigator, eralp çevikkalp, assoc prof, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bursa City Hospital 001
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Video-assisted Thoracoscopic Surgery (VATS); Serratus Posterior Superior Intercostal Plane Block
Keywords: Serratus posterior superior intercostal plane block; erector spinae plane block; pain management; Video-assisted thoracoscopic surgery (VATS)
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serratus posterior superior intercostal plane block (SPSIPB) (Active Comparator)
  Interventions: Other: Postoperative analgesia management(SPSIPB)
- Erector spinae plane block (Active Comparator)
  Interventions: Other: Postoperative analgesia management(ESPB)

INTERVENTIONS:
Other: Postoperative analgesia management(SPSIPB) — A high-frequency linear ultrasound probe (GE ML6-15-D Matrix Linear) will be covered with a sterile sheath, and the T3 level will be identified just above the medial border of the scapula. After visualizing the trapezius, rhomboid major, and serratus posterior superior muscles (from superficial to deep), 30 mL of 0.25% bupivacaine (Buvicaine 0.5%®, Polifarma, Tekirdağ, Türkiye) containing 7.5 µg epinephrine (1:200,000) (Adrenalin Bas Galen®; Galen, İstanbul, Türkiye) will be administered as the local anesthetic solution.
  Arms: Serratus posterior superior intercostal plane block (SPSIPB)
Other: Postoperative analgesia management(ESPB) — A high-frequency linear ultrasound probe (GE ML6-15-D Matrix Linear) will be covered with a sterile sheath. At the T5 vertebral level, the erector spinae muscle layers and the transverse process of the T5 vertebra, located immediately beneath them, will be identified. After confirming the transverse process, 30 mL of 0.25% bupivacaine (Buvicaine 0.5%®, Polifarma, Tekirdağ, Türkiye) containing 7.5 µg epinephrine (1:200,000) (Adrenalin Bas Galen®; Galen, İstanbul, Türkiye) will be administered as the local anesthetic solution.
  Arms: Erector spinae plane block

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) is a minimally invasive procedure performed through small thoracic incisions, but postoperative pain remains significant due to tissue and rib trauma. Poorly controlled pain may lead to chronic postoperative pain; therefore, optimal analgesia is essential.

According to PROSPECT guidelines, erector spinae plane block (ESPB) or paravertebral block (PVB) are recommended for VATS. The recently defined serratus posterior superior intercostal plane block (SPSIPB) provides analgesia between C3-T10 levels, but its efficacy compared with ESPB has not been studied.

This study aims to compare postoperative analgesic efficacy and patient satisfaction between ESPB and SPSIPB in VATS patients.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery (VATS) is a minimally invasive procedure performed through small thoracic incisions, but postoperative pain remains significant due to tissue and rib trauma. Poorly controlled pain may lead to chronic postoperative pain; therefore, optimal analgesia is essential.

According to PROSPECT guidelines, erector spinae plane block (ESPB) or paravertebral block (PVB) are recommended for VATS. The recently defined serratus posterior superior intercostal plane block (SPSIPB) provides analgesia between C3-T10 levels, but its efficacy compared with ESPB has not been studied.

This study aims to compare postoperative analgesic efficacy and patient satisfaction between ESPB and SPSIPB in VATS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years with ASA physical status I-III who will undergo elective video-assisted thoracoscopic surgery (VATS) will be included.

Exclusion Criteria:

* Patients who do not consent to participate in the study

Patients with coagulopathy

Patients with a history of local anesthetic allergy or toxicity

Patients with hepatic or renal failure

Patients with uncontrolled diabetes

Patients with uncontrolled hypertension

Mentally disabled patients

Patients receiving chronic pain treatment (opioid users)

Patients using antidepressant medication

Patients with neuropathic pain

Mentally disabled patients

Presence of infection at the injection site

Pregnant or breastfeeding women, or those with suspected pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | 0, 2, 4, 8, 16 and 24 hours
  Tramadol will be prepared as 5mg/ml and patient-controlled analgesia will be administered without basal infusion, with a locking time of 20 minutes and a bolus dose of 10mg.

SECONDARY OUTCOMES:
Postoperative pain scores (Numerical rating scale) (0-meaning "no pain" to 10-meaning "worst pain imaginable") | 0, 2, 4, 8, 16 and 24 hours
  Postoperative 24 hours period. Patients' pain scores will be questioned at 0, 2, 4, 8, 16 and 24 hours.
Global recovery scoring system (patient satisfaction scale)- QoR-15 | The quality of recovery will be evaluated out of a total of 150 points according to the QoR-15 test to be applied at the portoperative 24th hour.
  Researchers will use the Turkish version of the Quality Improvement Survey/QoR-15. PART A: Participants will be asked by researchers how they felt in the last 24 hours.(0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent]) 1. Able to breathe easily 2. Been able to enjoy food 3. Feeling rested 4. Have had a good sleep 5. Able to look after personal toilet and hygiene unaided 6. Able to communicate with 7. Getting support from hospital doctors and nurses 8. Able to return to work or usual home activities 9. Feeling comfortable and in control 10. Having a feeling of general well-being PART B Participants will be asked by the researchers whether they have experienced any of the following in the last 24 hours. (10 to 0, where: 10 = none of the time [excellent] and 0 = all of the time [poor]) 11. Moderate pain 12. Severe pain 13. Nausea or vomiting 14. Feeling worried or anxious 15. Feeling sad or depressed
Brief Pain Inventory | postoperative third month
  Brief Pain Inventory (BPI-Short Form) At the postoperative third month, patients will be contacted by phone, and chronic pain will be assessed using the Brief Pain Inventory - Short Form (BPI-SF).
  The BPI-SF consists of two main components:
  Pain Severity Score (0-10):
  Four numeric rating items evaluating worst, least, average, and current pain. Higher scores indicate more severe pain.
  Pain Interference Score (0-10):
  Seven numeric rating items evaluating interference with general activity, mood, walking ability, normal work, sleep, relations with others, and enjoyment of life.
  Higher scores indicate greater interference with daily activities.
Hospital Anxiety and Depression Scale (HADS) | On the morning of surgery and at the 3rd postoperative month
  The Hospital Anxiety and Depression Scale (HADS) was administered preoperatively and at the 3rd postoperative month. The change between these two time points will be included in the analysis.
  HADS consists of 14 items, divided into two subscales:
  HADS-Anxiety (HADS-A): 7 items
  HADS-Depression (HADS-D): 7 items
  Each item is scored on a 0-3 Likert scale, resulting in:
  HADS-A total score range: 0-21
  HADS-D total score range: 0-21
  Higher scores indicate worse anxiety or worse depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Mehta S, Jen TTH, Hamilton DL. Regional analgesia for acute pain relief after open thoracotomy and video-assisted thoracoscopic surgery. BJA Educ. 2023 Aug;23(8):295-303. doi: 10.1016/j.bjae.2023.05.001. Epub 2023 Jun 22. No abstract available. PMID 37465231
- [Background] Wong MKH, Sit AKY, Au TWK. Minimally invasive thoracic surgery: beyond surgical access. J Thorac Dis. 2018 Jun;10(Suppl 16):S1884-S1891. doi: 10.21037/jtd.2018.05.196. PMID 30026975
- [Background] Steinthorsdottir KJ, Wildgaard L, Hansen HJ, Petersen RH, Wildgaard K. Regional analgesia for video-assisted thoracic surgery: a systematic review. Eur J Cardiothorac Surg. 2014 Jun;45(6):959-66. doi: 10.1093/ejcts/ezt525. Epub 2013 Nov 27. PMID 24288340